CLINICAL TRIAL: NCT02345291
Title: A Phase 2a, Randomized, Double-blind, Placebo (Vehicle)-Controlled, Dose Finding Trial to Assess the Safety, Tolerability and Efficacy of NRD135S.E1 in Patients With Neuropathic Pain Associated With Diabetes Mellitus
Brief Title: Effect of NRD135S.E1 in Peripheral Neuropathic Pain in Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novaremed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NRD135S.E1-201
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-07

CONDITIONS: Diabetic Peripheral Neuropathic Pain
MeSH Terms: interventions — methyl N-acetylsibirosaminide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- NRD135S.E1 A (Experimental): A = 10 mg NRD135S.E1 once daily PO for 21 days
  Interventions: Drug: NRD135S.E1
- NRD135S.E1 B (Experimental): B = 40 mg NRD135S.E1 once daily PO for 21 days
  Interventions: Drug: NRD135S.E1
- NRD135S.E1 C (Experimental): C = 150 mg NRD135S.E1 once daily PO for 21 days
  Interventions: Drug: NRD135S.E1
- Placebo to match NRD135S.E1 D (Placebo Comparator): D = Placebo once daily PO for 21 days
  Interventions: Drug: Placebo to match NRD135S.E1

INTERVENTIONS:
Drug: NRD135S.E1 — A small chemical entity for treatment of neuropathic pain NRD135S.E1
  Other Names: E1
  Arms: NRD135S.E1 A; NRD135S.E1 B; NRD135S.E1 C
Drug: Placebo to match NRD135S.E1 — Placebo capsule to match NRD135S.E1 capsules
  Other Names: Placebo for E1
  Arms: Placebo to match NRD135S.E1 D

SUMMARY:
A multicenter, Phase 2a, randomized, double-blind, placebo (vehicle)-controlled, parallel-group, dose-finding study designed to evaluate the efficacy, safety and tolerability of NRD135S.E1 in adult patients with diabetes mellitus type 1 or 2 with neuropathic pain. Potential study patients will sign informed consent prior to undergoing any study-related procedure.

DETAILED DESCRIPTION:
Following screening, eligible patients will be enrolled and go through a week of washout of analgesic treatment. Patients who are still eligible following the washout will be randomized to one of four treatment groups: NRD135S.E1 at 10, 40, or 150 mg per day or placebo (vehicle).

All four treatment groups will start study treatment with 1 week of single blind placebo (baseline week) followed by 3 weeks of the allocated double blind treatment (Weeks 1, 2, and 3). All patients will be followed for 30 days after the last study drug administration. The total study duration per patient is 9 to10 weeks.

Visit schedule: Screening (Days minus 14 to minus 8, Visit 1). Washout visit (Day minus 7, Visit 2). Randomization and start of placebo treatment (Day 1, Visit 3). Double blind treatment visits on Days 8 (Visit 4), 15 (Visit 5) and 29 (Visit 6). Follow up visit by telephone (Day 59, Visit 7).

ELIGIBILITY:
Inclusion Criteria:

1. -Males agree to use condoms throughout treatment and follow up study periods.

   * Females must not be of childbearing potential as evidenced by at least one of the following:

     ≥ 62 years old and amenorrheic for ≥ 1 year
   * Amenorrheic ≥ 12 consecutive months and a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
   * Irregular menstrual periods and a documented FSH level > 35 mIU/mL
   * On hormone replacement therapy and prior clinical evidence of menopause based on any of the criteria above
   * Surgically sterile
2. Known stable diabetes mellitus for the last 3 months. (No oral hypoglycemic medications change allowed. Maximum insulin change allowed is ± 20%).
3. Evidence of peripheral neuropathy associated with diabetes mellitus diagnosed by DN4 criteria.
4. Presence of ongoing pain due to DPN for at least 3 months.
5. Mean DPN pain intensity of 4 to 9 on the NPS at screening.
6. HbA1c ≤ 9% of total hemoglobin at screening.
7. Willing to stop pain medications for DPN (except for limited use of paracetamol).
8. Signed written informed consent.

   * Subjects must have signed and dated an Institutional Review Board / Independent Ethics Committee approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
   * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.

Exclusion Criteria

1. Female of childbearing potential.
2. Neurologic disorders unrelated to DPN that may interfere with the assessment of DPN.
3. Known allergy or intolerance to paracetamol.
4. Evidence of non-DPN polyneuropathy.
5. The presence of severe pain associated with conditions other than DPN (e.g., peripheral vascular disease, phantom pain, etc.) that could confound the self-evaluation of pain due to DPN.
6. Any anti-epileptic or anti-depressive treatment. Amityptiline (Elatrol/Elatrolet) or duloxetine (Cymbalta) are permitted at screening but not later.
7. Constant use of non-steroidal anti-inflammatory drugs or opiates that cannot be withdrawn during the washout period and the whole study duration.
8. Participation in another clinical trial in the last 3 months.
9. Poor compliance with prescribed medication or alcohol or drug abuse within 2 years before screening.
10. Hypersensitivity to paracetamol or any of the inactive ingredients in NRD135S.E1 capsules.
11. Any serious medical condition, including the presence of laboratory abnormalities, that places the patient at an unacceptable risk if he or she participates in this study or confounds the ability to interpret data from the study.
12. Patients with any hematological disorder.
13. Prisoners or subjects who are involuntarily incarcerated.
14. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.
15. Patients whose judgment has been impaired by their physical ir mental condition

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
• Change from the baseline week to Week 3 in the weekly average daily pain intensity as measured on an 11-point numerical pain scale (NPS) | three weeks

SECONDARY OUTCOMES:
Change from the baseline week to Week 3 in the weekly maximum daily pain intensity as measured on the NPS | three weeks
Change from the baseline week to Week 3 in the weekly consumption of rescue analgesic (i.e., number of paracetamol 500 mg tablets taken per week) | three weeks
• Change from Day 8 (end of baseline week) to Day 29 (24 h after last study drug administration) in Short-Form McGill Pain Questionnaire (SF-MPQ) score | three
Clinician's Global Impression of Change from the baseline week at Day 29 (24 h after last study drug administration) | three weeks
Patient's Global Impression of Change from the baseline week at Day 29 (24 h after last study drug administration) | three weeks
Change from the baseline week to Week 3 in the weekly Daily Sleep Interference Score | three weeks
Incidence of treatment-emergent AEs (TEAEs) | three weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eli Kaplan, MD, Study Director — Novaremed Ltd.
Locations (10):
- Israel (10):
  - Diabetes and Endocrinology clinic, Bat-Yamon Medical center, Clalit health services, Bat Yam
  - Diabetes clinic, Lin Medical Center, Haifa
  - Rambam Medical Center, Diabetic Endocrine unit, Haifa
  - Wolfson Medical Center, Holon
  - Diabetic and Endocrinology clinic, Clalit health services, Jerusalem
  - Meir Medical Center, Endocrynology, diabetes and metabolism Unit, Kfar Saba
  - Ziv Medical Center, Endocrinology Unit, Safed
  - Diabetes Department Migdal Hamea Clalit health services, Tel Aviv
  - DMC Medical Center, Tel Aviv
  - Sorasky Medical Center, Diabetic unit, Tel Aviv

IPD SHARING:
Plan to Share IPD: Undecided